CLINICAL TRIAL: NCT00042731
Title: A Randomized Pilot Clinical Trial Of The Action Of Isoflavones And Lycopene In Localized Prostate Cancer: Administration Prior To Radical Prostatectomy
Brief Title: Isoflavones & Lycopene in Localized Prostate Ca:Prior to Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-13004; NCI-3811 (Other: NCI); NCI-P02-0216 (Other: NCI); 0105 (Other: CCOP)
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lycopene; Geritol; Soybean Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oral isoflavones with multivitamin (Active Comparator): Cohorts I - III: Patients receive 1 of 3 doses of oral isoflavones twice daily and a multivitamin once daily. Treatment in all arms continues for 4-6 weeks, until prostatectomy.
  Interventions: Dietary Supplement: Multivitamin; Dietary Supplement: Soy isoflavones
- Oral lycopene with multivitamin (Active Comparator): Cohorts IV-VI: Patients receive 1 of 3 doses of oral lycopene twice daily and a multivitamin once daily. Treatment in all arms continues for 4-6 weeks, until prostatectomy.
  Interventions: Dietary Supplement: Lycopene; Dietary Supplement: Multivitamin
- Multiple vitamin alone (Active Comparator): Patients receive a multivitamin once daily. Treatment in all arms continues for 4-6 weeks, until prostatectomy.
  Interventions: Dietary Supplement: Multivitamin

INTERVENTIONS:
Dietary Supplement: Lycopene — Daily administration as outlined in treatment arm(s)
  Arms: Oral lycopene with multivitamin
Dietary Supplement: Multivitamin — Daily administration as outlined in treatment arm(s)
Dietary Supplement: Soy isoflavones — Daily administration as outlined in treatment arm(s)
  Arms: Oral isoflavones with multivitamin

SUMMARY:
RATIONALE: Eating a diet rich in isoflavones, compounds found in soy foods, or lycopene, a substance found in tomatoes, may keep prostate cancer from growing. Giving isoflavones or lycopene before surgery may be an effective treatment for prostate cancer.

PURPOSE: Randomized clinical trial to compare the effectiveness of isoflavones with that of lycopene before surgery in treating patients who have stage I or stage II prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effect of isoflavones vs lycopene prior to radical prostatectomy on intermediate biomarkers (e.g., indices of cell proliferation and apoptosis) in patients with localized prostate cancer.
* Compare the effects of these nutritional supplements on increases in plasma levels and tissue levels of these agents in these patients.
* Compare the effects of these nutritional supplements on changes in surrogate markers of disease progression (e.g., prostate-specific antigen levels) in these patients.
* Compare the effects of these nutritional supplements on changes in serum steroid hormones, estradiol, and free testosterone in these patients.
* Compare the magnitude of these changes in patients treated with these nutritional supplements vs patients in the control group.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease stage (stage I vs stage II) and presence of high-grade prostatic intraepithelial neoplasia. Patients are randomized to 1 of 7 treatment groups.

PROJECTED ACCRUAL: A total of 87 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed localized prostate cancer

  * Stage I or II
* Scheduled prostatectomy between 4-6 weeks after initial biopsy

PATIENT CHARACTERISTICS:

Age:

* 45 to 80

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* No known history of hepatic disease

Renal:

* No known history of renal disease

Other:

* No known history of thyroid disease
* Body mass index no greater than 32
* Omnivorous diet
* No known allergy to study supplements
* No evidence of prostatitis or urinary tract infection
* No other prior malignancy except nonmelanoma skin cancer
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* No concurrent thyroid hormone replacement medications

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Other:

* At least 30 days since prior antibiotics
* At least 30 days since prior diet high in soy and/or lycopene products (e.g., greater than 40 mg soy/day and/or greater than 15 mg lycopene/day)
* No other concurrent nutritional supplements, including modular supplements with other carotenoids and isoflavones
* No prior or concurrent therapy for prostate cancer

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2002-07; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Occurrences of Treatment Effect on Biomarkers in Each Group | 4 years
  Effect of isoflavones and lycopene on endpoint biomarkers as measured by tissue cell proliferation, apoptosis, or programmed cell death at prostate cancer biopsy and surgical excision

SECONDARY OUTCOMES:
Occurrences of Plasma Level Changes for Each Group | 4 years
  Plasma levels of isoflavones and lycopene as measured by plasma analysis at baseline and post-study intervention
Occurrence of Tissue Level Increases | 4 years
  Correlation of plasma and tissue levels of isoflavones and lycopene as measured by plasma and tissue analysis at baseline and post-study intervention
Occurrences of Disease Progression for Each Group | 4 years
  Effect of isoflavones and lycopene on markers of disease progression as measured by prostate-specific antigen (PSA) levels at baseline and post-study intervention
Occurrences of Hormonal Effect | 4 years
  Effect of isoflavones and lycopene on serum steroid hormones as measured by sex-hormone-binding globulin, estradiol, and free testosterone at baseline and post-study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nagi B. Kumar, PhD, RD, FADA, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (5):
- United States (5):
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - CCOP - Scott and White Hospital, Temple, Texas